CLINICAL TRIAL: NCT03564769
Title: Evaluation Study of SPOTme® Skin Cancer Screenings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: American Academy of Dermatology (AAD) (Unknown)
Responsible Party: Principal Investigator, Alan Geller, MPH, RN, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17-1668
Record Dates: First submitted 2017-12-06; First posted 2018-06-21 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Skin Cancer
Keywords: screening
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm 1 (Experimental): Individuals randomized to intervention group 1 will have participated in the AAD SPOTmeⓇ skin cancer screening program in either 2016 or 2017 AND will receive additional skin cancer screening educational materials.
  Interventions: Behavioral: Intervention Arm; Other: AAD SPOTmeⓇ skin cancer screening
- Intervention Arm 2 (Experimental): Individuals randomized to intervention group 2 will have participated in the AAD SPOTmeⓇ skin cancer screening program in either 2016 or 2017 only.
  Interventions: Other: AAD SPOTmeⓇ skin cancer screening

INTERVENTIONS:
Behavioral: Intervention Arm — Individuals randomized to the intervention group will receive skin cancer screening educational materials.
  Arms: Intervention Arm 1
Other: AAD SPOTmeⓇ skin cancer screening — All study participants will have participated in the AAD SPOTmeⓇ skin cancer screening program in either 2016 or 2017.

SUMMARY:
This study evaluates the impact of the AAD SPOTme® skin cancer screening events on attendees' skin cancer prevention and detection behaviors. This study will also evaluate whether an educational intervention will improve post-screening engagement of attendees with dermatologists.

DETAILED DESCRIPTION:
Despite tremendous growth in both the interest and volume of skin cancer screenings at the national level, the actual utility and impact of the AAD SPOT me™ skin cancer screening programs have not been fully evaluated. This study will address this knowledge gap. Early detection is vital in the fight against skin cancer, the most common cancer in the United States. While the effects of skin cancer can be devastating, this disease is highly treatable when detected early.

This study evaluates the impact of the AAD SPOTme® skin cancer screening events on attendees' skin cancer prevention and detection behaviors. This study will also evaluate whether an educational intervention will improve post-screening engagement of attendees with dermatologists.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the American Academy of Dermatology national screening program in 2016 or 2017
* Have a presumptive diagnosis (screening, non-confirmed) of melanoma
* Have provided the AAD with permission to be re-contacted
* Have provided the AAD with an email address
* Aged 18 years or older
* Able to read English

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Completion of a physician skin examination | Baseline
  Self-report of a physician skin examination will be defined as a health care provider examining the patient's entire body for any sign of skin cancer during the period following patient's receipt of an AAD SPOTme® skin cancer screening to the baseline assessment.

SECONDARY OUTCOMES:
Completion of a physician skin examination | 6 months
  Self-report of a physician skin examination will be defined as a health care provider examining the patient's entire body for any sign of skin cancer during the 3 months prior to the 6-month follow up assessment
Patient thorough skin self-examination (TSSE) | 6 months
  Self-report of patient thorough skin self-examination (TSSE) will be defined as performing at least one TSSE during the 3 months prior to the 6-month follow up assessment
Patient attitude towards sun protection | 6 months
  Self-report of patient attitude towards use of sun protection will be defined by likelihood of engaging in sun protection practices in the year following the 6-month follow up assessment

CONTACTS AND LOCATIONS:
Overall Officials: Alan Geller, MPH, RN, Principal Investigator — Harvard TH Chan School of Public Health
Locations (1):
- Harvard TH Chan School of Public Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No